CLINICAL TRIAL: NCT00694733
Title: Regulation of Cortisol Metabolism and Fat Patterning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jonathan Purnell, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: eIRB #937; OCTRI #862 (Other: Oregon Health and Sciences University)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Menopausal Syndrome
Keywords: Obesity; Menopausal Syndrome; Cortisol
MeSH Terms: conditions — Obesity | interventions — Saline Solution; Aromatase Inhibitors; Testosterone; Gels; Anastrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Men on placebo injections for 4 months
  Interventions: Drug: Placebo injection
- 2 (Active Comparator): Men who receive Depo Lupron for 4 months, then are replaced with testosterone and aromatase inhibitor for 4 months.
  Interventions: Drug: Depo Lupron/Aromatase inhibitor
- 3 (Active Comparator): Men who receive Depo Lupron for 4 months, then are replaced with testosterone and placebo for 4 months.
  Interventions: Drug: Depo Lupron/placebo
- 4 (Placebo Comparator): Women on placebo cream
  Interventions: Drug: placebo
- 5 (Active Comparator): Women on estrogen cream
  Interventions: Drug: Estrogen cream

INTERVENTIONS:
Drug: Placebo injection — Normal saline injection IM monthly for 4 months
  Other Names: Normal Saline
  Arms: 1
Drug: Depo Lupron/Aromatase inhibitor — Depo Lupron injection 7.5mg IM monthly for 8 months, with addition of testosterone gel and aromatase inhibitor months 4-8.
  Other Names: Depo-Lupron; Testim 1% gel; Anastrozole; Arimidex
  Arms: 2
Drug: Depo Lupron/placebo — Depo Lupron injection 7.5mg IM monthly for 8 months, with addition of testosterone gel and placebo months 4-8.
  Other Names: Depo-Lupron; Testim 1% gel; Placebo capsules
  Arms: 3
Drug: placebo — Placebo Cream 1ml applied twice daily for four months
  Other Names: Placebo cream
  Arms: 4
Drug: Estrogen cream — Estrogen cream 1 ml twice daily, dose titrated to maintain estradiol level between 60 and 280 pg/ml.
  Other Names: Estradiol cream
  Arms: 5

SUMMARY:
The purpose of this study is to determine if estrogen or testosterone can affect cortisol levels and where fat builds up in our bodies.

DETAILED DESCRIPTION:
Subjects will be studied 3 or 4 times on the inpatient unit of the Oregon Clinical and Translational Research Center. During each visit, testing will include measuring the amount of whole body fat and fat in the stomach area, muscle, and liver; levels of cortisol in the blood, urine, and fat tissue (taken from a biopsy); how well insulin works (insulin sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* 40 postmenopausal women (age 40-62) and 30 men (age 18-45) will be recruited if they are healthy, at their lifetime maximal weight, have been weight stable for at least six months prior to entry, have a BMI between 19 and 39.9 kg/m2, and be willing to commit to not making significant changes to their diet or daily activities while enrolled in the study.

Exclusion Criteria:

* Subjects will be excluded for potential confounders on body weight, cortisol production rates, sex steroid metabolism, or contraindications to strong magnetic fields:

  1. Age less than 18 to exclude those who might be experiencing alterations in cortisol production or weight as a result of adolescent growth
  2. Subjects who exercise > 30 minutes/day, 3 times a week
  3. Smokers
  4. Heavy alcohol drinkers (> 2 drinks/ day)
  5. Subjects with medical diagnosis including diabetes, heart disease, and cancer
  6. Subjects with psychiatric illness (i.e., depression, psychosis, bipolar, schizophrenia; or are taking medications for these disorders)
  7. BMI 40 kg/m2, since obesity influences levels of sex steroids and sex hormone binding globulin; or body weight > 136 kg (300 lbs), since this is the weight limit for the DEXA and MR machines
  8. Presence of metal in the body such as body piercing, shrapnel, cardiac pacemakers or aneurysm clips
  9. Endocrine diseases affecting body composition, such as untreated hypothyroidism or Cushing's syndrome, will be excluded by history and physical examination, or by laboratory evaluation if necessary.
* Women with a contraindication to estrogen use will also be excluded, including: an estrogen dependent malignancy, active thrombophlebitis, history of deep venous thrombosis, hypertriglyceridemia, untreated hypertension, cardiovascular disease, migraine headaches, or current tobacco use.
* Women with frequent hot flashes or disrupted sleep will also be excluded since they will be unlikely to tolerate randomization to placebo and continued symptoms and altered sleep cycles will independently affect cortisol secretion patterns.
* All volunteers will have had a normal mammogram within the previous 12 months.
* Any subject with previously unevaluated postmenopausal bleeding will not be included and, instead, will be referred to a physician for evaluation.
* Women who underwent surgical menopause (bilateral ovariectomy) must be at least one year out from their surgery before considered eligible so as to allow weight stabilization after the procedure.
* Men will have had a prostate exam by their primary health provider within the previous year or by the PI at the time of screening for this study.
* Any subjects taking a blood thinning medication or with an abnormal exam will not be included and, instead, will be referred to a physician for evaluation

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2005-05; Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
To measure 24-hour CPR, free cortisol, and cortisol binding globulin levels in plasma; HSD 1 activity, glucocorticoid receptor binding, and cortisol levels in adipocytes; and urinary excretion of cortisol, cortisone and their metabolites. | Before and after hormone replacement therapy

SECONDARY OUTCOMES:
To measure intramyocellular fat and intrahepatic fat by MRS, visceral and subcutaneous abdominal fat by CT scan, body composition (fat mass, lean mass, and bone mass) by DXA, and insulin sensitivity. | Before and after hormone replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, M.D., Principal Investigator — OHSU - Center for the Study of Weight Regulation
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States